CLINICAL TRIAL: NCT01002625
Title: Double-Blind, Randomized, Multiple-Dose, Placebo-Controlled, 2-Way Crossover Study To Study Effects Of PF-04457845 On Polysomnographic Endpoints In Healthy Volunteers
Brief Title: A Study To Establish The Effects Of PF-04457845 On Sleep In Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: B0541008
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2010-07

CONDITIONS: Sleep; Healthy Volunteers
Keywords: Double-Blind Randomized Placebo-Controlled 2-Way Crossover Polysomnographic Endpoints
MeSH Terms: interventions — N-pyridazin-3-yl-4-(3-((5-(trifluoromethyl)pyridin-2-yl)oxy)benzylidene)piperidine-1-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. PF-04457845 followed by placebo (Experimental): PF-04457845 followed by placebo
  Interventions: Drug: PF-04457845 / matched placebo
- 2. Placebo followed by PF-04457845 (Experimental): Placebo followed by PF-04457845
  Interventions: Drug: PF-04457845 / matched placebo

INTERVENTIONS:
Drug: PF-04457845 / matched placebo — PF-04457845 4 mg tablet once daily / matched placebo
  Arms: 1. PF-04457845 followed by placebo
Drug: PF-04457845 / matched placebo — PF-04457845 4 mg tablet once daily / matched placebo
  Arms: 2. Placebo followed by PF-04457845

SUMMARY:
PF-04457845 has been shown to temporarily decrease the dream (REM) period of sleep in rats, which suggests that PF-04457845 is active in rat's brains. This study is designed to see whether this is also the case in man.

DETAILED DESCRIPTION:
The trial was terminated prematurely December 3, 2009 owing to an operational error. There were no safety or efficacy concerns relating to the study and the decision to terminate the trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years Body Mass Index (BMI) between 17.5 and 30.5 kg/m2; and a total body weight >50 kg

Exclusion Criteria:

* History of any active sleep disorder.
* History of any sleep or circadian rhythm sleep disorder including RLS, narcolepsy, sleep apnea, phase advance or delay syndromes within the past 5 years.
* Currently on or planning to be involved in night or rotating shift work or traveling across more than four time zones in 14 days prior to screening.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Percentage of total sleep time spent in REM (ie, time spent in REM/total sleep time * 100). | 3 days

SECONDARY OUTCOMES:
Percentage of total sleep time spent in Stage 1 sleep | 3 days
Percentage of total sleep time spent in Stage 2 sleep | 3 days
Percentage of total sleep time spent in Stage 3-4 sleep | 3 days
Total sleep time | 3 days
Sleep efficiency (total sleep time/time in bed * 100). | 3 days
Wake after sleep onset (sum of wake time during sleep and prior to final awakening) and wake time after sleep) (WASO). | 3 days
Number of arousals after sleep onset (NASO | 3 days
Latency to persistent sleep | 3 days
Plasma concentrations of PF-04457845. | 3 days
Plasma concentrations of fatty acid amides. | 3 days
Beta-band spectral power (qEEG) measured with eyes open and eyes closed while subjects are awake immediately before lights off for each PSG. | 3 days
Beta-band spectral power (qEEG) measured with eyes open and eyes closed while subjects are awake immediately after lights on for each PSG. | 3 days
Beta-band spectral power (qEEG) measured while subjects are asleep during the sleep onset period (SOP) and first 3 periods of NREM sleep. | 3 days
For definitions of polysomnography variable objectives and endpoints see Appendix 3 | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New York, New York, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0541008&StudyName=A%20Study%20To%20Establish%20The%20Effects%20Of%20PF-04457845%20On%20Sleep%20In%20Healthy%20Volunteers